CLINICAL TRIAL: NCT02964260
Title: Randomized Controlled Trial of Transarterial Embolization Simultaneously Combined Thermal Ablation for Large Hepatocellular Carcinoma
Brief Title: RCT of TAE Simultaneously Combined Thermal Ablation for Large Hepatocellular Carcinoma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Collaborators: First Affiliated Hospital, Sun Yat-Sen University (Other); Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other); Third Affiliated Hospital, Sun Yat-Sen University (Other); Sixth Affiliated Hospital, Sun Yat-sen University (Other); Guangdong Provincial People's Hospital (Other)
Responsible Party: Principal Investigator, Huang Jinhua, Professor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TASAL
Record Dates: First submitted 2016-11-09; First posted 2016-11-16 (Estimated); Last update posted 2021-05-14 (Actual); Status verified 2021-05

CONDITIONS: Hepatocellular Carcinoma, Adult
Keywords: HCC; Embolization; Ablation; simultaneously; sequentially
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Drug Therapy; Embolization, Therapeutic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- TAE combined ablation simultaneously (Experimental): TAE simultaneously combined with ablation.The treatment interval is 1-3 days between two procedures. TAE using embolic agents(Lipiodol/Gelatin sponge/PVA particles(300～500μm)/Blank microspheres).
  Interventions: Drug: Embolic agents; Procedure: Simultaneously; Device: Ablation
- TACE combined ablation sequentially (Other): TACE sequentially combined thermal ablation.The treatment interval is 1 month between two procedures. TACE using chemotherapy drug(Doxorubicin/platinum agents) and embolic agents(Lipiodol/Gelatin sponge/PVA particles(300～500μm)/Blank microspheres).
  Interventions: Drug: Chemotherapy drug; Drug: Embolic agents; Procedure: Sequentially; Device: Ablation

INTERVENTIONS:
Drug: Chemotherapy drug — Doxorubicin/Platinum agents
  Other Names: Chemotherapy
  Arms: TACE combined ablation sequentially
Drug: Embolic agents — Lipiodol/Gelatin sponge/PVA/Blank microspheres
  Other Names: Embolization
Procedure: Simultaneously — 1-3 days
  Other Names: Treatment interval
  Arms: TAE combined ablation simultaneously
Procedure: Sequentially — 1 month
  Other Names: Treatment interval
  Arms: TACE combined ablation sequentially
Device: Ablation — Radiofrequency ablation/Microwave ablation
  Other Names: RFA/MWA

SUMMARY:
This study intends to evaluate the efficacy and safety of Transarterial embolization (TAE) simultaneously combined with thermal ablation for large hepatocellular carcinoma (HCC). Half participants will receive TAE simultaneously combined with thermal ablation and the other half receive TACE sequentially combined with thermal ablation, which is a conventional treatment for HCC patients.

DETAILED DESCRIPTION:
The treatment method "Transarterial chemoembolization (TACE) sequentially combined with thermal ablation" is recommend for large HCC patients from NCCN Guideline and Chinese guideline "Diagnosis and Treatment of Primary Liver Cancer". The details of this sequential method consist one or more times of TACE followed by thermal ablation at least one month later to make the tumor completely inactivate. The thermal ablations include multiple applicators radiofrequency or microwave ablations. However, this method includes such disadvantages. 1) The limitation of lipiodol dosage in one TACE session is 30ml so that many patients needs more sessions of TACE; (2) Lipiodol and chemical drugs is easy to leak when patients have hepatic arteriovenous fistula. (3) Repeated TACE could cause more serious side effects. (4) Tumors of many patients are still not controlled or grow too large to ablate after TACEs which increases the metastasis risk and affects the efficacy and survival time.

However, TAE simultaneously combined with thermal ablation is another combination type which reduce the interval time between two procedures from one month to 1-3 days. TAE removes the chemical drugs and uses embolic agents such as Embosphere to obstruct vessels to enhance the effect of followed ablations. The main aim of reducing interval and remove chemical drugs is to make the tumor completely inactivate in one hospitalization like surgical operation, hoping bringing less side effects, better efficacy and longer survival time.

Thus the investigators will launch a prospective, multicenter randomized controlled clinical trial to compare the 3-years overall survival, safety, social and economic benefit of TAE simultaneously combined with ablation and TACE sequentially combined with ablation. The investigators expect to acquire Ia-level evidence-based medical evidence which can be accepted by the clinical guideline, popularizing, demonstrating our therapy.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 to 70 years with estimated survival over 3 months
* Number of tumors < 3
* Diameter of tumor between 5cm to 15cm
* No portal vein trunk tumoral thrombus or inferior vena cava tumoral thrombus
* With arteriovenous fistula or arterioportal shunt fistula that can be completely embolized
* Child-Pugh class A or B/Child score > 7;ECOG score < 2
* Tolerable coagulation function or reversible coagulation disorders
* Laboratory examination test: WBC≥3.0×10E9/L; Hb≥3.0×10E9/L; PLT ≥50×10E9/L; INR < 2.3 or PT< 16.5s; Cr ≤ 145.5 umul/L
* Signed informed consent before recruiting

Exclusion Criteria:

* Diffused HCC
* With portal vein trunk tumoral thrombus
* With inferior vena cava tumoral thrombus or hepatic vein tumor thrombus
* With lymphatic metastasis or extra hepatic metastasis
* Child-Pugh class C and can't be improved by expectant treatment
* Untreatable coagulation disorders, severe hemogram abnormal and bleeding tendency
* Massive intractable ascites
* ECOG score > 2

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 410 (Estimated)
Dates: Start 2016-05 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Overall survival | 3 years
  From complete remission of the index large tumor to patient death or the completion of this trial

SECONDARY OUTCOMES:
Recurrence free survival | 3 years
  From complete remission of the index large tumor to tumor recurrence either in- or extra- hepatic or the completion of this trial
liver and renal function | 3 years
  Alanine aminotransferase,Ast,total bilirubin,albumin,creatinine,Urea nitrogen
Complications | 3 years
  number of participants with Complications
Times of interventional procedures | 3 years
  The number of procedures for each patient, either TACE/TAE or ablation

CONTACTS AND LOCATIONS:
Overall Officials: Jinhua Huang, Ph.D, Principal Investigator — Sun Yat-sen University
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No